CLINICAL TRIAL: NCT02190357
Title: Rifaximin Reduces the Complications of Decompensated Cirrhosis
Brief Title: Rifaximin Reduces the Complications of Decompensated Cirrhosis: a Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPDLCC-2
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Cirrhosis
Keywords: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rifaximin (Experimental): 400 mg bid,orally
  Interventions: Drug: Rifaximin
- controlled group (No Intervention): no intervention

INTERVENTIONS:
Drug: Rifaximin — Rifaximin is an antibiotic that is virtually non-absorbed after oral administration and exhibits broad spectrum antimicrobial activity against both aerobic and anaerobic gram-positive and gram-negative microorganisms within the gastrointestinal tract.
  Arms: rifaximin

SUMMARY:
Cirrhotic patients are predisposed to intestinal dysmotility, bacterial overgrowth, and increased intestinal permeability all leading to an increase in bacterial translocation and increased endotoxemia. Rifaximin is an antibiotic that is virtually non-absorbed after oral administration and exhibits broad spectrum antimicrobial activity against both aerobic and anaerobic gram-positive and gram-negative microorganisms within the gastrointestinal tract. It has been suggested that oral prophylactic antibiotics or bowel decontamination might improve long-term outcomes in patients with cirrhosis. The aim of this study was to explore the effect of rifaximin on the complications of advanced cirrhosis.

DETAILED DESCRIPTION:
Cirrhotic patients are predisposed to intestinal dysmotility, bacterial overgrowth, and increased intestinal permeability all leading to an increase in bacterial translocation and increased endotoxemia. Cirrhotics with bacterial translocation and endotoxemia manifest hemodynamic derangement with lower systemic vascular resistance, higher cardiac output, and lower mean arterial pressure. Moreover, endotoxins may increase portal pressure by increasing vascular resistance which may be promoted through the cytokine-stimulated intrahepatic release of endothelin and cyclo-oxygenase products.

Indeed, bacterial infections are common in cirrhotic patients and have approximately 30% mortality at one month and a further 30% mortality at 12 months as documented in a systematic review comprising almost 12 000 patients. It follows that altering gut flora to decrease endotoxin levels may lead to improved prognosis in cirrhosis. Rifaximin is an antibiotic that is virtually non-absorbed after oral administration and exhibits broad spectrum antimicrobial activity against both aerobic and anaerobic gram-positive and gram-negative microorganisms within the gastrointestinal tract. It has been suggested that oral prophylactic antibiotics or bowel decontamination might improve long-term outcomes in patients with cirrhosis, not only by reducing the risk of infections but also by reducing hepatic vein pressure gradient (HVPG).

The aim of this study was to explore the effect of rifaximin on the complications of advanced cirrhosis.

ELIGIBILITY:
1. Eligicility criteria (1) Willing to give written informed consent and comply with the study restrictions and requirements (2) Age from 18 to 75 years at screening (3) Clinical diagnosis of decompensated liver cirrhosis
2. Exclusion criteria (1) Episodes of overt hepatic encephalopathy (HE), esophageal gastric variceal bleeding (EGVB) or spontaneous bacterial peritonitis (SBP) within one month (2) Hepatitis B Virus (HBV) DNA ≥ 500 copy/ml (3) Standard antiviral treament duration less than six months for patients receiving antiviral treatment for hepatitis B or hepatitis C (4) Planned to receive or change the antiviral treament projects at the screening (5) Unwilling to stop alcohol abuse after inclusion (≥20 g/ d for women or ≥40 g/d for men) (6) Serum total bilirubin ≥ 170 μmol/L (7) Serum sodium level < 125 mmol/L (8) White blood cell count < 1×109/L (9) Serum creatinine ≥ 1.2 fold of upper limits of normal (10) Clinically diagnosed or suspected as liver malignancy (11) Previous use of antibiotics within two weeks before inclusion (12) HIV seropositivity (13) Poorly controlled hypertension, diabetes mellitus or other severe heart and lung diseases (14) Known hypersensitivity to rifaximin (15) Pregnancy and lactation woman (16) Participated in other studies within three months before screening (17) Not suitble for participating the study judged by investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
number of death | 6 months
numbers of liver transplantation | 6 months
numbers of hepatic encephalopathy | 6 months
Numbers of other complications of cirrhosis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Xie, MD, Principal Investigator — Department of Gastroenterology, Changzheng Hospital, Second Military Medical University, Shanghai
Locations (1):
- Shanghai changzheng Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Mullen KD, Sanyal AJ, Bass NM, Poordad FF, Sheikh MY, Frederick RT, Bortey E, Forbes WP. Rifaximin is safe and well tolerated for long-term maintenance of remission from overt hepatic encephalopathy. Clin Gastroenterol Hepatol. 2014 Aug;12(8):1390-7.e2. doi: 10.1016/j.cgh.2013.12.021. Epub 2013 Dec 21. PMID 24365449
- [Result] Xu D, Gao J, Gillilland M 3rd, Wu X, Song I, Kao JY, Owyang C. Rifaximin alters intestinal bacteria and prevents stress-induced gut inflammation and visceral hyperalgesia in rats. Gastroenterology. 2014 Feb;146(2):484-96.e4. doi: 10.1053/j.gastro.2013.10.026. Epub 2013 Oct 22. PMID 24161699
- [Result] Lutz P, Parcina M, Bekeredjian-Ding I, Hoerauf A, Strassburg CP, Spengler U. Spontaneous bacterial peritonitis by Pasteurella multocida under treatment with rifaximin. Infection. 2014 Feb;42(1):175-7. doi: 10.1007/s15010-013-0449-4. Epub 2013 Mar 25. PMID 23526308
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180
- [Derived] Zeng X, Sheng X, Wang PQ, Xin HG, Guo YB, Lin Y, Zhong JW, He CZ, Yin J, Liu TT, Ma WJ, Xiao X, Shi PM, Yuan ZL, Yang L, Ma X, Xu JM, Shen XZ, Yang CQ, Zhu X, Lv NH, Xie WF. Low-dose rifaximin prevents complications and improves survival in patients with decompensated liver cirrhosis. Hepatol Int. 2021 Feb;15(1):155-165. doi: 10.1007/s12072-020-10117-y. Epub 2021 Jan 1. PMID 33385299